CLINICAL TRIAL: NCT02590887
Title: Clinical Study to Assess the Immunomodulatory and Antioxidant Effects of a Beverage Manufactured From Lupine Protein Hydrolysates in Healthy Volunteers
Brief Title: Safety and Efficacy of a Drink Containing Lupine Protein Hydrolysates on the Immune, Oxidative and Metabolic Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Antonio Carrillo Vico, PhD, University of Seville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Lupine-1
Record Dates: First submitted 2015-10-22; First posted 2015-10-29 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Healthy Volunteers

ARMS (1):
- drink manufactured from lupine peptides (Experimental): Beverage drink containing 0.5mg/ml of protein hydrolysate extracted from food grade lupine flour. The drink will be formulated as 200 mL tetra brik subjected to a test of microbiological safety according to the Spanish law (RD 135/2010 of 12 February 2010).
  The final beverage shall consist of:
  * Oily phase: refined sunflower oil 5% w/w of the emulsion
  * Aqueous phase (water) 95% w/w of the emulsion, containing equal volumes of solution A and B:
    * Solution A:
      * Hydrolyzed Lupine (1.17% w/w)
      * Sucrose (14.03% w/w)
      * Vanilla flavor (0.42% w/w)
      * Drinking water (84.38% w/v)
    * Solution B:
      * Xanthan gum (0.28% w/w)
      * Drinking water (99.72% w/v)
  The samples will guard and kept by the investigator until the day of delivery to the volunteers.
  The duration of treatment 4 weeks, during which the volunteers daily consume the contents of a tetra brik.
  Interventions: Dietary Supplement: Drink manufactured from lupine peptides

INTERVENTIONS:
Dietary Supplement: Drink manufactured from lupine peptides — Comparison of blood levels of immune, oxidative stress, biochemical markers and haemogram before and after (14, and 28 days) drinking the beverage.

SUMMARY:
The purpose of this study is to determine the health effects of the 4 weeks daily intake of a drink manufactured from lupine protein hydrolysates in healthy volunteers. For that, blood markers of inflammation, oxidative stress, carbohydrate, lipid, protein and liver metabolism, together with general hematology and blood coagulation will be assessed at baseline time (day 0) and after drink ingestion (day +14 and +28).

DETAILED DESCRIPTION:
The main objective of the present study is to verify the hypothesis that the intake of the drink based on lupine peptides is safe and has beneficial effects on the immune and oxidative status.

The secondary objectives are:

* Assess the effect of the drink on biological parameters of the carbohydrate, lipid, renal and hepatic metabolism as well as hematology analysis.
* Assess whether the new product is well tolerated.
* Evaluate the effect of the drink on the general health of the volunteers through the Short Form-36 health survey.
* Determine the degree of drink acceptability through the acceptability Likert test.

ELIGIBILITY:
Inclusion Criteria:

* Subject between 18 and 50 years old
* Body mass index between 19 and 26 kg/m2
* No severe disease
* Biochemical markers within the normal range
* No previous history of drug abuse
* Negative serology for hepatitis C virus (HCV), hepatitis B virus (HBV) and HIV
* Females must have a negative pregnancy test
* The volunteer should signed the informed consent approved by the Ethics Committees of Clinical Trials

Exclusion Criteria:

* Pre-existing disease
* Treatment with anti-inflammatory, antipyretic or antibiotic drugs
* Smoker
* Harmful alcohol consumption according to World Health Organization standards
* Pregnant females
* Hypersensitivity to lupine, corn or xanthan gum.
* Allergies to plant derivatives and celiac.
* Participation in another clinical trial.
* Blood donation in the previous three months.
* Any other circumstance that according to the research team may lead to increased risk for voluntary

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Assessment of the change from baseline of the plasma total antioxidant activity | day 0 (baseline), +14, +28, +42
  Plasma total antioxidant activity
Assessment of the change from baseline of the plasma superoxide dismutase activity | day 0 (baseline), +14, +28, +42
  Plasma superoxide dismutase activity
Assessment of the change from baseline of the plasma catalase activity | day 0 (baseline), +14, +28, +42
  Plasma catalase activity
Assessment of the change from baseline of the plasma gluthathione peroxidase activity | day 0 (baseline), +14, +28, +42
  Plasma gluthathione peroxidase activity
Assessment of the change from baseline of the plasma gluthathione reductase activity | day 0 (baseline), +14, +28, +42
  Plasma gluthathione reductase activity
Assessment of the change from baseline of the plasma levels of C reactive protein | day 0 (baseline), +14, +28, +42
  Plasma levels of C reactive protein
Assessment of the change from baseline of the plasma levels of immunoglobulins | day 0 (baseline), +14, +28, +42
  plasma levels of immunoglobulin A, immunoglobulin E, immunoglobulin G and immunoglobulin M
Assessment of the change from baseline of the plasma levels of complement | day 0 (baseline), +14, +28, +42
  plasma levels of C3 and C4
Assessment of the change from baseline of the cytokines production in peripheral blood mononuclear cells | day 0 (baseline), +14, +28, +42
  Supernatant levels of Interleukin (IL-1)beta, IL-2, IL-4, IL-5, IL-6, IL-9, IL-10, IL-12, IL-13, IL-17, IL-22, IFNgamma and Tumour necrosis factor (TNF)-alpha

SECONDARY OUTCOMES:
Assessment of the change from baseline of the plasma levels of glucose | day 0 (baseline), +14, +28, +42
  Plasma levels of glucose
Assessment of the change from baseline of haematological markers | day 0 (baseline), +14, +28, +42
  Haemogram
Assessment of the change from baseline of the plasma levels of homocysteine | day 0 (baseline), +14, +28, +42
  Plasma levels of homocysteine
Assessment of the change from baseline of the plasma levels of insulin | day 0 (baseline), +14, +28, +42
  Plasma levels of insulin
Assessment of the change from baseline of the plasma levels of triglycerides | day 0 (baseline), +14, +28, +42
  Plasma levels of triglycerides
Assessment of the change from baseline of the plasma levels of cholesterol | day 0 (baseline), +14, +28, +42
  Plasma levels of cholesterol
Assessment of the change from baseline of the plasma levels of Low Density Lipoprotein (LDL) cholesterol | day 0 (baseline), +14, +28, +42
  Plasma levels of LDL cholesterol
Assessment of the change from baseline of the plasma levels of High Density Lipoprotein (HDL) cholesterol | day 0 (baseline), +14, +28, +42
  Plasma levels of HDL cholesterol
Assessment of the change from baseline of the plasma levels of total proteins | day 0 (baseline), +14, +28, +42
  Plasma levels of total proteins
Assessment of the change from baseline of the plasma levels of urea | day 0 (baseline), +14, +28, +42
  Plasma levels of urea
Assessment of the change from baseline of the plasma levels of creatinine | day 0 (baseline), +14, +28, +42
  Plasma levels of creatinine
Assessment of the change from baseline of the plasma levels of alkaline phosphatase | day 0 (baseline), +14, +28, +42
  Plasma levels of alkaline phosphatase
Assessment of the change from baseline of the plasma levels of Alanine Aminotransferase (ALT) | day 0 (baseline), +14, +28, +42
  Plasma levels of ALT
Assessment of the change from baseline of the plasma levels of Aspartate Aminotransferase (AST) | day 0 (baseline), +14, +28, +42
  plasma levels of AST
Assessment of the change from baseline of the plasma levels of Gamma-Glutamyltransferase (GGT) | day 0 (baseline), +14, +28, +42
  plasma levels of GGT
Assessment of the change from baseline of the gene expression of antioxidant enzymes in peripheral blood mononuclear cells | day 0 (baseline), +14, +28, +42
  Messenger Ribonucleic Acid (mRNA) expression of superoxide dismutase, Catalase, Gluthathione peroxidase, Gluthathione reductase and inducible nitric oxide synthase (iNOS)
Assessment of the change from baseline of the Body Mass Index | day 0 (baseline), +14, +28, +42
  Body Mass Index

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carrillo Vico, PhD, Principal Investigator — University of Seville
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Spain

REFERENCES:
- [Background] Millan-Linares Mdel C, Yust Mdel M, Alcaide-Hidalgo JM, Millan F, Pedroche J. Lupine protein hydrolysates inhibit enzymes involved in the inflammatory pathway. Food Chem. 2014 May 15;151:141-7. doi: 10.1016/j.foodchem.2013.11.053. Epub 2013 Nov 19. PMID 24423513
- [Background] Cruz-Chamorro I, Alvarez-Sanchez N, Millan-Linares MDC, Yust MDM, Pedroche J, Millan F, Lardone PJ, Carrera-Sanchez C, Guerrero JM, Carrillo-Vico A. Lupine protein hydrolysates decrease the inflammatory response and improve the oxidative status in human peripheral lymphocytes. Food Res Int. 2019 Dec;126:108585. doi: 10.1016/j.foodres.2019.108585. Epub 2019 Jul 27. PMID 31732051